CLINICAL TRIAL: NCT04077112
Title: Evaluation of Intensive Parent-Child Interaction Therapy"
Acronym: IPCIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-16-0323-CR03
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Behavior Problem; Parenting
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional PCIT (Active Comparator): once a week parent training
  Interventions: Behavioral: Parent Child Interaction Therapy
- intensive PCIT (Experimental): every day for two weeks parent training
  Interventions: Behavioral: Parent Child Interaction Therapy

INTERVENTIONS:
Behavioral: Parent Child Interaction Therapy — Behavioral parent training program targeting parent-child relationship

SUMMARY:
The purpose to the current study was to examine the comparative efficacy of a more condensed intensive version of Parent-Child Interaction Therapy (I-PCIT; 5 days/week over the course of 2 weeks) versus a more traditional weekly PCIT format (1 day/week over the course of 10 weeks) in treating early childhood externalizing behavior problems (EBP).

DETAILED DESCRIPTION:
The purpose to the current study was to examine the comparative efficacy of a more condensed intensive version of Parent-Child Interaction Therapy (I-PCIT; 5 days/week over the course of 2 weeks) versus a more traditional weekly PCIT format (1 day/week over the course of 10 weeks) in treating early childhood externalizing behavior problems (EBP). Using a randomized trial design, 60 young children (M child age = 4.33 years; range 2-6.92; 65% male; 85% Latinx) with elevated levels of EBP and their mothers were assigned to either I-PCIT (n = 30) or traditional PCIT (n = 30). Families completed pre-treatment and post-treatment assessments as well as a follow-up assessment 6-9 months following treatment completion. Across all assessments, mothers completed measures of child behavior, discipline practices, and parenting stress. Observational data on child behavior and parenting was also collected during three 5-minute standard situations that vary in the degree of parental control (child-led play, parent-led play, & clean-up).

ELIGIBILITY:
Inclusion Criteria:

* children had to be between 2 and 7 years of age
* mothers had to rate their children above the clinically significant range (T-score > 60) on a measure of child EBP (Eyberg Child Behavior Inventory; Eyberg & Pincus, 1999),
* be willing to come to treatment every day (Monday - Friday) during a two-week period,
* both mother and child had to be able to speak and understand English.

Exclusion Criteria:

* An intellectual disability (full scale IQ < 70 based on the WPPSI-IV; Wechsler, 2012),
* A previous Autism Spectrum Disorder diagnosis,
* The inability of parents to attend sessions daily.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Externalizing Behavior Problems | The measure was collected prior to the start of treatment, immediately following treatment, as well as 6-9 months upon treatment completion
  Mothers completed the Eyberg Child Behavior Inventory (ECBI; Eyberg & Ross, 1978), a 36-item questionnaire that is designed to assess the presence of externalizing problems in children ages 2 through 16 years. The total intensity scale t-score was used in the current study as the main measure of EBP (α's .84-.93).
  The total raw score ranged from 36 to 252. Higher scores indicate the presence of more externalizing behavior problems.

SECONDARY OUTCOMES:
Change in Parenting Skills | The measure was collected prior to the start of treatment, immediately following treatment, as well as 6-9 months upon treatment completion
  The Dyadic Parent-Child Interaction Coding System-4th Edition (DPICS-IV; Eyberg, Nelson, Ginn, Bhuiyan, & Boggs, 2013), an established behavioral coding system was used to measure the quality of parent-child interactions across all assessments. Consistent with prior PCIT research, we created a composite of do skills (behavior descriptions, reflections, praises) and don't skills (questions, commands, and negative talk) reflecting behaviors parents are taught during treatment to use and not use during a child-led play. Undergraduate student coders, who were masked to treatment status, were trained to 80% agreement with a criterion tape and coded 20% of the observations a second time to assess reliability. Reliability for the do (r's range from .87 to .94) and don't skills were excellent (r's .99).
Change in Parenting stress | The measure was collected prior to the start of treatment, immediately following treatment, as well as 6-9 months upon treatment completion
  Mothers completed the Parenting Stress Index-Short Form (PSI-SF; Abidin, 1983). The PSI-SF is a widely used 36-item self-report instrument for parents of children ages 1 month to 12 years measuring parental stress (Abidin, 1983). The PSI-SF total raw score was used to measure overall parenting stress (α's .88-.94). Total score range from 36 to 180 with higher scores indicating greater levels of parenting stress.
Change in Discipline Practices | The measure was collected prior to the start of treatment, immediately following treatment, as well as 6-9 months upon treatment completion
  Mothers completed the Parenting Scale (PS; Arnold, O'Leary, Wolff, & Acker, 1993), a 30-item self-report measure that assesses parental discipline practices of children as young as 18 months. The effectiveness of discipline techniques is measured based on three factor scores (Laxness, Over-Reactivity, Verbosity). The Laxness (α's = .82-.88) and Over-Reactivity (α's = .67-.83) scales were used to assess parenting practices. Due to poor reliability of the Verbosity scale (.33-.70), this scale was removed from all analyses.

IPD SHARING:
Plan to Share IPD: No
final data set will be available upon request